CLINICAL TRIAL: NCT03682120
Title: A Phase II Study in Healthy Adults 18-64 Years Old to Assess the Safety, Reactogenicity and Immunogenicity of a Seqirus A/H7N9 Inactivated Influenza Vaccine Administered Intramuscularly With or Without MF59(R) Adjuvant
Brief Title: Safety/Efficacy Study of Seqirus A/H7N9 IIV With or Without MF59(R) Adjuvant to Prevent Avian Influenza
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-0076; HHSN272201300021I
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Results first posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2018-09-13

CONDITIONS: Avian Influenza; Influenza Immunisation
Keywords: A/H7N9; Healthy Adults; Immunogenicity; Influenza vaccine; MF59(R) adjuvant; Reactogenicity; Safety
MeSH Terms: conditions — Influenza in Birds; Influenza, Human | interventions — MF59 oil emulsion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 (Experimental): 3.75 mcg per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + MF59(R) adjuvant administered intramuscularly on Day 1 and Day 22. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages. N=106
  Interventions: Biological: A/H7N9; Drug: MF59; Other: Phosphate Buffered Saline (PBS) diluent
- Arm 2 (Experimental): 7.5 mcg per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + MF59(R) adjuvant administered intramuscularly on Day 1 and Day 22. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages. N=106
  Interventions: Biological: A/H7N9; Drug: MF59; Other: Phosphate Buffered Saline (PBS) diluent
- Arm 3 (Experimental): 15 mcg per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + MF59(R) adjuvant administered intramuscularly on Day 1 and Day 22. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages. N=106
  Interventions: Biological: A/H7N9; Drug: MF59; Other: Phosphate Buffered Saline (PBS) diluent
- Arm 4 (Experimental): 15 mcg per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) unadjuvanted administered intramuscularly on Day 1 and Day 22. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages. N=53
  Interventions: Biological: A/H7N9; Other: Phosphate Buffered Saline (PBS) diluent

INTERVENTIONS:
Biological: A/H7N9 — Monovalent inactivated, "subunit" influenza virus vaccine containing the HA and NA from influenza A/Hong Kong/125/2017 (H7N9) and the PB2, PB1, PA, NP, M and NS genes from A/Puerto Rico/8/1934 (H1N1).
Drug: MF59 — Microfluoridized adjuvant 59 (MF59) is an oil-in-water emulsion.
  Arms: Arm 1; Arm 2; Arm 3
Other: Phosphate Buffered Saline (PBS) diluent — Diluent for Influenza Virus Vaccine.

SUMMARY:
This is a randomized, double-blinded, Phase II study in healthy males and non-pregnant females, 18-64 years of age. This clinical trial is designed to assess the safety, reactogenicity, and immunogenicity of a pre-pandemic 2017 monovalent inactivated influenza A/H7N9 virus vaccine (2017 H7N9 IIV) manufactured by Seqirus Inc (Seqirus) administered at different dosages (3.75 microgram mcg, 7.5 mcg and 15 mcg of hemagglutinin (HA) per dose) given with MF59(R) adjuvant manufactured by Seqirus Inc., or without adjuvant (15 mcg of HA per dose). Phosphate buffered saline (PBS) diluent manufactured by Patheon Manufacturing Services LLC will be used to achieve certain targeted doses. Approximately 371 subjects who are in good health and meet all eligibility criteria will be randomized into one of 4 study groups. The study will be conducted at up to 7 Vaccine and Treatment Unit (VTEU) sites and will last approximately 17 months, with subject participation duration of approximately 13 months. The Primary Objectives of the study are: 1) To assess the safety and reactogenicity following receipt of two doses of 2017 H7N9 IIV administered intramuscularly (IM) at different dosages approximately 21 days apart given with or without MF59(R) adjuvant; 2) To assess the serum hemagglutinin inhibition (HAI) and neutralizing (Neut) antibody responses approximately 21 days following receipt of two doses of 2017 H7N9 IIV administered IM at different dosages approximately 21 days apart with or without MF59(R) adjuvant.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, Phase II study in healthy males and non-pregnant females, 18-64 years of age. This clinical trial is designed to assess the safety, reactogenicity, and immunogenicity of a pre-pandemic 2017 monovalent inactivated influenza A/H7N9 virus vaccine (2017 H7N9 IIV) manufactured by Seqirus Inc (Seqirus) administered at different dosages (3.75 mcg, 7.5 mcg and 15 mcg of hemagglutinin (HA) per dose) given with MF59(R) adjuvant manufactured by Seqirus Inc., or without adjuvant (15 mcg of HA per dose). Phosphate buffered saline (PBS) diluent manufactured by Patheon Manufacturing Services LLC will be used to achieve certain targeted doses. Approximately 371 subjects who are in good health and meet all eligibility criteria will be randomized into one of 4 study groups. The study will be conducted at up to 7 Vaccine and Treatment Unit (VTEU) sites and will last approximately 17 months, with subject participation duration of approximately 13 months. The Primary Objectives of the study are: 1) To assess the safety and reactogenicity following receipt of two doses of 2017 H7N9 IIV administered intramuscularly (IM) at different dosages approximately 21 days apart given with or without MF59(R) adjuvant; 2) To assess the serum hemagglutinin inhibition (HAI) and Neutralizing (Neut) antibody responses approximately 21 days following receipt of two doses of 2017 H7N9 IIV administered IM at different dosages approximately 21 days apart with or without MF59(R) adjuvant.

The secondary Objectives are: 1) To assess all unsolicited non-serious Adverse Events (AEs) following receipt of two doses of a 2017 H7N9 IIV administered IM at different dosages approximately 21 days apart with or without MF59(R) adjuvant; 2) To assess medically-attended adverse events (MAAEs) including new-onset chronic medical conditions (NOCMCs), potentially immune-mediated medical conditions (PIMMCs), and all Serious Adverse Events (SAEs) following receipt of two doses of a 2017 H7N9 IIV administered IM at different dosages approximately 21 days apart with or without MF59(R) adjuvant; 3) To assess the serum HAI and Neut antibody responses approximately 7 and 21 days following receipt of a single dose, and approximately 7 days following receipt of two doses of 2017 H7N9 IIV administered IM at different dosages approximately 21 days apart with or without MF59(R) adjuvant.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Are males or non-pregnant females, 18-64 years of age, inclusive.
4. Are in good health*. *As determined by physical examination and medical history to evaluate acute or currently ongoing chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days, which would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days (no hospitalizations, Emergency Room, or urgent care for condition and no adverse symptoms that need medical intervention such as medication change/supplemental oxygen). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided there was no deterioration in the subject's chronic medical condition that necessitated a medication change, and there is no additional risk to the subject or interference with the evaluation of responses to study vaccination. [Topical, nasal, and inhaled medications (with the exception of inhaled corticosteroids), herbals, vitamins, and supplements are permitted].
5. Oral temperature is less than 100.0 degree Fahrenheit.
6. Pulse is 47 to 100 beats per minute, inclusive.
7. Systolic blood pressure is 85 to 150 millimeters of Mercury, inclusive.
8. Diastolic blood pressure is 55 to 95 millimeters of Mercury, inclusive.
9. Women of childbearing potential* must agree to practice an acceptable contraception method** from 30 days before first study vaccination until 60 days after last study vaccination.

   *Not sterilized via tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or < 1 year of the last menses if menopausal.

   **Includes non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving the first study vaccination, barrier methods such as male or female condoms with spermicide or with the use of applied spermicide, intrauterine devices, NuvaRing(R), and licensed hormonal methods such as implants, injectables, or oral contraceptives ("the pill").
10. Women of childbearing potential must have a negative serum or urine pregnancy test within 24 hours prior to study vaccination.

Exclusion Criteria:

1. Have an acute illness*, as determined by the site Principal Investigatoor or appropriate sub-investigator, within 72 hours prior to study vaccination.

   *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site principal investigator or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
2. Have any medical disease or condition that, in the opinion of the site Principal Investigator or appropriate sub-investigator, is a contraindication to study participation*.

   *Including acute or chronic medical disease or condition, defined as persisting for at least 90 days, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
3. Have immunosuppression as a result of an underlying illness or treatment, a recent history or current use of immunosuppressive or immunomodulating disease therapy.
4. Use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
5. Have known active neoplastic disease or a history of any hematologic malignancy. Non-melanoma, treated, skin cancers are permitted.
6. Have known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection.
7. Have known hypersensitivity or allergy to eggs, egg or chicken protein, neomycin, kanamycin, formaldehyde, polysorbate 80, cetyltrimethylammonium bromide (CTAB), squalene-based adjuvants, or other components of the study vaccine.
8. Have a history of severe reactions following previous immunization with licensed or unlicensed influenza vaccines.
9. Have a history of Guillian-Barre Syndrome.
10. Have a history of convulsions or encephalomyelitis within 90 days prior to study vaccination.
11. Have a history of Potentially Immune Mediated Medical Conditions (PIMMCs)
12. Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
13. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
14. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
15. Have taken oral or parenteral (including intra-articular) corticosteroids of any dose within 30 days prior to study vaccination.
16. Have taken high-dose inhaled corticosteroids* within 30 days prior to each study vaccination.

    *High-dose defined as per age as using inhaled high dose per reference chart https://www.nhlbi.nih.gov/files/docs/guidelines/asthma_qrg.pdf.
17. Received a licensed live vaccine within 30 days prior to the first study vaccination, or plan to receive a licensed live vaccine within 30 days before or after each study vaccination.
18. Received or plan to receive a licensed, inactivated, vaccine (excluding all flu vaccines) within 14 days before or after each study vaccination.
19. Received or plan to receive seasonal inactivated influenza virus (IIV) within 21 days before or after each study vaccination.
20. Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within 90 days prior to each study vaccination.
21. Received an experimental agent* within 30 days prior to the first study vaccination, or expect to receive an experimental agent** during the 13-month trial-reporting period.

    *Including vaccine, drug, biologic, device, blood product, or medication.

    **Other than from participation in this trial.
22. Are participating or plan to participate in another clinical trial with an interventional agent* that will be received during the 13-month trial-reporting period.

    *Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.
23. Received or plan to receive an influenza A / H7 vaccine* or have a history of influenza A / H7 subtype infection.

    *And assigned to a group receiving influenza A / H7 vaccine, does not apply to documented placebo recipients.
24. Have traveled to mainland China and had substantial* direct contact with live or freshly slaughtered poultry or pigeons within the past five years.

    *Substantial contact is defined as visited a poultry farm and/or a live poultry market.
25. Occupational exposure to or substantial direct physical contact* with birds in the past year and through the 21 days after the second study vaccination.

    *Exposure to free range chickens in the yard is exclusionary. Casual contact with birds at petting zoos or county or state fairs or having pet birds does not exclude subjects from study participation.
26. Female subjects who are breastfeeding at any given time from the first study vaccination until 30 days after the last study vaccination.
27. Plan to travel outside the US (continental US, Hawaii, and Alaska) from enrollment through 21 days after the second study vaccination.
28. Receipt of Multimeric-001 (M-001) vaccine.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 372 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Alabama at Birmingham School of Medicine - Alabama Vaccine Research Clinic, Birmingham, Alabama
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Vanderbilt University Medical Center - Vanderbilt Institute for Clinical and Translational Research - Clinical Research Center (VICTR-CRC), Nashville, Tennessee
  - The University of Texas Medical Branch - Sealy Center for Vaccine Development (SCVD), Galveston, Texas
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - Kaiser Permanente Washington Health Research Institute - Vaccines and Infectious Diseases, Seattle, Washington

REFERENCES:
- [Derived] Frey SE, Brady R, Jackson L, Goepfert P, El Sahly HM, Atmar RL, Rupp R, Creech CB, Abate G, Paulsen G, Weiss J, Wegel A, Roberts PC. Safety and immunogenicity of ascending doses of influenza A(H7N9) inactivated vaccine with or without MF59(R). Vaccine. 2025 Feb 15;47:126702. doi: 10.1016/j.vaccine.2024.126702. Epub 2025 Jan 10. PMID 39798434

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy males and non-pregnant females between 18 and 64 years old, inclusively. They were recruited from the communities at large around the clinical sites. Participants were enrolled between 27NOV2018 and 02APR2019.
Groups:
- 3.75 mcg A/H7N9+MF59: 3.75 mcg per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + MF59(R) adjuvant administered intramuscularly on Day 1 and Day 22. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  A/H7N9: Monovalent inactivated, "subunit" influenza virus vaccine containing the HA and NA from influenza A/Hong Kong/125/2017 (H7N9) and the PB2, PB1, PA, NP, M and NS genes from A/Puerto Rico/8/1934 (H1N1).
  MF59 adjuvant: Microfluoridized adjuvant 59 (MF59) is an oil-in-water emulsion.
  Phosphate Buffered Saline (PBS) diluent: Diluent for Influenza Virus Vaccine.
- 7.5 mcg A/H7N9+MF59: 7.5 mcg per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + MF59(R) adjuvant administered intramuscularly on Day 1 and Day 22. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  A/H7N9: Monovalent inactivated, "subunit" influenza virus vaccine containing the HA and NA from influenza A/Hong Kong/125/2017 (H7N9) and the PB2, PB1, PA, NP, M and NS genes from A/Puerto Rico/8/1934 (H1N1).
  MF59 adjuvant: Microfluoridized adjuvant 59 (MF59) is an oil-in-water emulsion.
  Phosphate Buffered Saline (PBS) diluent: Diluent for Influenza Virus Vaccine.
- 15 mcg A/H7N9+MF59: 15 mcg per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + MF59(R) adjuvant administered intramuscularly on Day 1 and Day 22. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  A/H7N9: Monovalent inactivated, "subunit" influenza virus vaccine containing the HA and NA from influenza A/Hong Kong/125/2017 (H7N9) and the PB2, PB1, PA, NP, M and NS genes from A/Puerto Rico/8/1934 (H1N1).
  MF59 adjuvant: Microfluoridized adjuvant 59 (MF59) is an oil-in-water emulsion.
  Phosphate Buffered Saline (PBS) diluent: Diluent for Influenza Virus Vaccine.
- 15 mcg A/H7N9: 15 mcg per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) unadjuvanted administered intramuscularly on Day 1 and Day 22. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  A/H7N9: Monovalent inactivated, "subunit" influenza virus vaccine containing the HA and NA from influenza A/Hong Kong/125/2017 (H7N9) and the PB2, PB1, PA, NP, M and NS genes from A/Puerto Rico/8/1934 (H1N1).
  Phosphate Buffered Saline (PBS) diluent: Diluent for Influenza Virus Vaccine.
Period: Overall Study
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Started | 105 | 105 | 105 | 57
Completed | 92 | 97 | 97 | 55
Not Completed | 13 | 8 | 8 | 2
Not completed — Lost to Follow-up | 11 | 4 | 5 | 2
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 3 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Enrolled but Treatment Not Administered | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all enrolled participants
Groups:
- 3.75 mcg A/H7N9+MF59: 3.75 mcg per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + MF59(R) adjuvant administered intramuscularly on Day 1 and Day 22. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
- 7.5 mcg A/H7N9+MF59: 7.5 mcg per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + MF59(R) adjuvant administered intramuscularly on Day 1 and Day 22. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
- 15 mcg A/H7N9+MF59: 15 mcg per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + MF59(R) adjuvant administered intramuscularly on Day 1 and Day 22. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
- 15 mcg A/H7N9: 15 mcg per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) unadjuvanted administered intramuscularly on Day 1 and Day 22. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
- Total: Total of all reporting groups
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9 | Total
Number analyzed (Participants) | 105 | 105 | 105 | 57 | 372
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 105 | 105 | 105 | 57 | 372
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (13.6) | 40.5 (13.7) | 38.8 (13.3) | 43.8 (15.1) | 40.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 63 | 65 | 29 | 216
  Male | 46 | 42 | 40 | 28 | 156
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 10 | 3 | 26
  Not Hispanic or Latino | 98 | 99 | 95 | 54 | 346
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 7 | 6 | 3 | 4 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 17 | 12 | 16 | 13 | 58
  White | 78 | 81 | 82 | 37 | 278
  More than one race | 2 | 4 | 2 | 2 | 10
  Unknown or Not Reported | 1 | 2 | 2 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 105 | 105 | 105 | 57 | 372
Prior Seasonal Influenza Vaccination (2017-2018 or 2018-2019) [Count of Participants; unit: Participants]
  Neither | 17 | 18 | 23 | 14 | 72
  2017-2018 Only | 10 | 8 | 8 | 4 | 30
  2018-2019 Only | 17 | 14 | 14 | 6 | 51
  Both 2017-2018 and 2018-2019 | 61 | 65 | 60 | 33 | 219

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMT) of Serum Hemagglutinin Inhibition (HAI) Antibodies
Description: Blood was collected for HAI assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 21 days after the second dose of H7N9 (Day 43).
Time Frame: Day 43
Population: The modified intent-to-treat (mITT) population includes all participants who received at least one study vaccination and contributed both pre- and at least one post-study vaccination venous blood samples for HAI antibody assays for which valid results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 102 | 101 | 101 | 55
titer | 23.3 [17.9 to 30.3] | 19.9 [15.8 to 25.1] | 24.2 [18.8 to 31.1] | 6.0 [5.6 to 6.6]

2. Primary Outcome: Geometric Mean Titers (GMT) of Serum Neutralizing (Neut) Antibodies
Description: Blood was collected for Neutralizing assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 21 days after the second dose of H7N9 (Day 43).
Time Frame: Day 43
Population: The modified intent-to-treat (mITT) population includes all participants who received at least one study vaccination and contributed both pre- and at least one post-study vaccination venous blood samples for Neut antibody assays for which valid results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 102 | 101 | 101 | 55
titer | 24.9 [20.1 to 30.7] | 24.1 [19.6 to 29.6] | 28.0 [22.8 to 34.4] | 6.4 [5.6 to 7.2]

3. Primary Outcome: Number of Participants With Clinical Safety Laboratory Adverse Events
Description: Laboratory parameters include alanine aminotransferase (ALT), bilirubin, creatinine, hemoglobin, platelets and white blood cells (WBC). Thresholds for adverse events were considered as ALT 44 IU/L or greater (female) or 61 IU/L or greater (male); bilirubin 1.30 mg/dL or greater; creatinine 1.1 mg/dL or greater (female) or 1.4 mg/dL or greater (male); hemoglobin 11.4 g/dL or lower (female) or 12.4 g/dL or lower (male); platelets 139 x10^3/µL or below or 416 x10^3/µL or greater; or WBC or 3.9 x10^3/µL or lower or 10.6 x10^3/µL or higher.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine. Participants with at least one lab result reported for Day 8 were included for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- 7.5 mcg A/H7N9: 15 mcg per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) unadjuvanted administered intramuscularly on Day 1 and Day 22. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9
Number analyzed (Participants) | 105 | 104 | 102 | 57
Participants
  WBC | 9 | 8 | 5 | 2
  Hemoglobin | 4 | 5 | 2 | 4
  Platelets | 2 | 3 | 5 | 0
  ALT | 3 | 1 | 1 | 0
  Total Bilirubin | 0 | 1 | 1 | 1
  Creatinine | 4 | 0 | 1 | 1

4. Primary Outcome: Number of Participants With Clinical Safety Laboratory Adverse Events
Description: as for outcome 3
Time Frame: Day 22 to Day 29
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine. Participants with at least one lab result reported for Day 29 were included for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 96 | 96 | 95 | 53
Participants
  WBC | 11 | 13 | 9 | 4
  Hemoglobin | 3 | 6 | 2 | 1
  Platelets | 3 | 6 | 0 | 0
  ALT | 2 | 2 | 1 | 0
  Total Bilirubin | 1 | 1 | 1 | 2
  Creatinine | 1 | 1 | 1 | 0

5. Primary Outcome: Number of Participants With Solicited Injection Site Reactogenicity Events
Description: Injection site AEs solicited on a memory aid provided to participants included Pain, Tenderness, Itching/Pruritus, Ecchymosis/Bruising (functional grade based on interference with daily activities), Ecchymosis/Bruising (any measured value >0mm), Erythema/Redness (functional grade), Erythema/ Redness (any measured value >0mm), Induration/Swelling (functional grade), and Induration/Swelling (any measured value >0mm). Participants are considered reporting the injection site AE if they reported mild or greater severity at any time during the 8 days at or following the first vaccination.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine. Participants who received the first dose of study vaccine were included for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 105 | 104 | 57
Participants | 78 | 76 | 70 | 20

6. Primary Outcome: Number of Participants With Solicited Injection Site Reactogenicity Events
Description: Injection site AEs solicited on a memory aid provided to participants included Pain, Tenderness, Itching/Pruritus, Ecchymosis/Bruising (functional grade based on interference with daily activities), Ecchymosis/Bruising (any measured value >0mm), Erythema/Redness (functional grade), Erythema/ Redness (any measured value >0mm), Induration/Swelling (functional grade), and Induration/Swelling (any measured value >0mm). Participants are considered reporting the injection site AE if they reported mild or greater severity at any time during the 8 days at or following the second vaccination.
Time Frame: Day 22 through Day 29
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine. Participants who received the second dose of study vaccine were included for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 97 | 99 | 97 | 54
Participants | 63 | 55 | 57 | 13

7. Primary Outcome: Number of Participants With Study Vaccine-related Serious Adverse Events (SAEs)
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect. Events are included if deemed by the investigator to be related to the study product.
Time Frame: Day 1 through Day 387
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 105 | 104 | 57
Participants | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Systemic Reactogenicity Events
Description: Systemic AEs solicited on a memory aid provided to participants included Elevated Oral Temperature, Feverishness, Fatigue, Malaise, Myalgia, Arthralgia, Headache, and Nausea. Participants are considered reporting the systemic AE if they reported mild or greater severity at any time during the 8 days at or following the first vaccination.
Time Frame: Day 1 through Day 8
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 105 | 104 | 57
Participants | 50 | 43 | 39 | 23

9. Primary Outcome: Number of Participants With Systemic Reactogenicity Events
Description: Systemic AEs solicited on a memory aid provided to participants included Elevated Oral Temperature, Feverishness, Fatigue, Malaise, Myalgia, Arthralgia, Headache, and Nausea. Participants are considered reporting the systemic AE if they reported mild or greater severity at any time during the 8 days at or following the second vaccination.
Time Frame: Day 22 through Day 29
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 97 | 99 | 97 | 54
Participants | 29 | 37 | 27 | 9

10. Primary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study group from the available results at 21 days after second dose of H7N9 (Day 43).
Time Frame: Day 43
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 102 | 101 | 101 | 55
percentage of participants | 43 [33 to 53] | 30 [21 to 40] | 40 [30 to 50] | 0 [0 to 6]

11. Primary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Titers of 1:40 or Greater
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study group from the available results at 21 days after second dose of H7N9 (Day 43).
Time Frame: Day 43
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 102 | 101 | 101 | 55
percentage of participants | 45 [35 to 55] | 42 [32 to 52] | 44 [34 to 54] | 2 [0 to 10]

12. Primary Outcome: Percentage of Participants Achieving Seroconversion Defined by Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 21 days after second dose of H7N9 is Day 43.
Time Frame: Day 43
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 102 | 101 | 101 | 55
percentage of participants | 43 [33 to 53] | 30 [21 to 40] | 40 [30 to 50] | 0 [0 to 6]

13. Primary Outcome: Percentage of Participants Achieving Seroconversion Defined by Neutralizing (Neut) Antibodies
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 21 days after second dose of H7N9 is Day 43.
Time Frame: Day 43
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 102 | 101 | 101 | 55
percentage of participants | 45 [35 to 55] | 42 [32 to 52] | 44 [34 to 54] | 2 [0 to 10]

14. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for HAI assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at baseline (Day 1).
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 103 | 103 | 57
titer | 5.3 [5.1 to 5.4] | 5.3 [5.1 to 5.6] | 5.3 [5.2 to 5.5] | 5.3 [5.1 to 5.6]

15. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for HAI assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 7 days post first vaccination (Day 8).
Time Frame: Day 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 103 | 103 | 56
titer | 5.4 [5.2 to 5.5] | 5.4 [5.2 to 5.6] | 6.0 [5.5 to 6.5] | 6.2 [5.0 to 7.7]

16. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for HAI assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 21 days post first vaccination (Day 22).
Time Frame: Day 22
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 104 | 102 | 102 | 56
titer | 6.1 [5.5 to 6.6] | 5.8 [5.5 to 6.1] | 7.5 [6.5 to 8.7] | 6.1 [4.9 to 7.6]

17. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for HAI assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 7 days post second vaccination (Day 29).
Time Frame: Day 29
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 96 | 97 | 97 | 54
titer | 17.4 [13.4 to 22.5] | 15.9 [12.6 to 20.1] | 23.6 [18.5 to 30.0] | 6.5 [5.5 to 7.3]

18. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Neutralizing (Neut) Antibodies
Description: Blood was collected for Neutralizing assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at baseline (Day 1).
Time Frame: Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 103 | 103 | 57
titer | 5.0 [5.0 to 5.1] | 5.0 [5.0 to 5.1] | 5.1 [5.0 to 5.1] | 5.0 [5.0 to 5.0]

19. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Neutralizing (Neut) Antibodies
Description: Blood was collected for Neutralizing assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 7 days post first vaccination (Day 8).
Time Frame: Day 8
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 103 | 103 | 56
titer | 5.2 [5.1 to 5.3] | 5.2 [5.1 to 5.4] | 5.5 [5.2 to 5.8] | 5.1 [5.0 to 5.3]

20. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Neutralizing (Neut) Antibodies
Description: Blood was collected for Neutralizing assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 21 days post first vaccination (Day 22).
Time Frame: Day 22
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 104 | 102 | 102 | 56
titer | 6.3 [5.8 to 6.8] | 6.1 [5.6 to 6.6] | 7.0 [6.4 to 7.7] | 5.2 [5.0 to 5.4]

21. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Neutralizing (Neut) Antibodies
Description: Blood was collected for Neutralizing assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 7 days post second vaccination (Day 29).
Time Frame: Day 29
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 96 | 97 | 97 | 54
titer | 19.2 [15.8 to 23.3] | 18.9 [15.4 to 23.1] | 25.2 [20.6 to 30.9] | 6.3 [5.6 to 7.0]

22. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Regardless of the Assessment of Relatedness
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect. All events are included regardless of relationship to the study product.
Time Frame: Day 1 through Day 387
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 105 | 104 | 57
Participants | 1 | 6 | 4 | 1

23. Secondary Outcome: Number of Participants With Unsolicited Adverse Events, Regardless of the Assessment of Seriousness or Relatedness
Description: Adverse events were defined as any untoward medical occurrence in a participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Non-serious AEs were collected from participants at follow up visits through 21 days after each vaccination. Adverse events were MedDRA coded and are summarized by MedDRA System Organ Class (SOC).
Time Frame: Day 1 through Day 22
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine. Participants who received Vaccination 1 were included for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 105 | 104 | 57
Participants | 23 | 22 | 27 | 14

24. Secondary Outcome: Number of Participants With Unsolicited Adverse Events, Regardless of the Assessment of Seriousness or Relatedness
Description: as for outcome 23
Time Frame: Day 22 through Day 43
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine. Participants who received Vaccination 2 were included for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- 3.75 mcg A/H7N9+MF596: 3.75 mcg per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + MF59(R) adjuvant administered intramuscularly on Day 1 and Day 22. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
Arm/Group | 3.75 mcg A/H7N9+MF596 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 97 | 99 | 97 | 54
Participants | 19 | 18 | 18 | 14

25. Secondary Outcome: Number of Participants With Medically-Attended Adverse Events (MAAEs), New-Onset Chronic Medical Conditions (NOCMCs), and Potentially Immune-Mediated Medical Conditions (PIMMCs)
Description: Participants were queried at each visit for the occurrence of medically-attended adverse events (MAAEs), including new-onset chronic medical conditions (NOCMCs) and potentially immune-mediated medical conditions (PIMMCs) throughout the duration of the study.
Time Frame: Day 1 through Day 387
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 105 | 104 | 57
Participants
  Medically-attended adverse events | 23 | 35 | 35 | 18
  New onset chronic medical condition | 6 | 7 | 6 | 2
  Potentially immune-mediated medical condition | 0 | 0 | 1 | 0

26. Secondary Outcome: Number of Participants With Study Vaccine-related Unsolicited Non-serious Adverse Events (AEs)
Description: Adverse events were defined as any untoward medical occurrence in a participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Non-serious AEs were collected from participants at follow up visits through 21 days after each vaccination. The site investigator determined vaccine related as "a reasonable possibility that the study product caused the AE. Reasonable possibility means that there is evidence to suggest a causal relationship between the study product and the AE." Adverse events were MedDRA coded and are summarized by MedDRA System Organ Class (SOC).
Time Frame: Day 1 through Day 22
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 105 | 104 | 57
Participants | 9 | 5 | 5 | 2

27. Secondary Outcome: Number of Participants With Study Vaccine-related Unsolicited Non-serious Adverse Events (AEs)
Description: as for outcome 26
Time Frame: Day 22 through Day 43
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 97 | 99 | 97 | 54
Participants | 5 | 4 | 5 | 3

28. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study group from the available results at baseline (Day 1).
Time Frame: Day 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 103 | 103 | 57
percentage of participants | 0 [0 to 3] | 0 [0 to 4] | 0 [0 to 4] | 0 [0 to 6]

29. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study group from the available results at 7 days post first vaccination (Day 8).
Time Frame: Day 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 103 | 103 | 56
percentage of participants | 0 [0 to 3] | 0 [0 to 4] | 2 [0 to 7] | 4 [0 to 12]

30. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study group from the available results at 21 days post first vaccination (Day 22).
Time Frame: Day 22
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 104 | 102 | 102 | 56
percentage of participants | 4 [1 to 10] | 0 [0 to 4] | 6 [2 to 12] | 4 [0 to 12]

31. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study group from the available results at 7 days post second vaccination (Day 29).
Time Frame: Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 96 | 97 | 97 | 54
percentage of participants | 34 [25 to 45] | 26 [17 to 36] | 40 [30 to 51] | 2 [0 to 10]

32. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Titer of 1:40 or Greater
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of subjects with Neut titer >= 1:40 was calculated for each study group from the available results at baseline (Day 1).
Time Frame: Day 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 103 | 103 | 57
percentage of participants | 0 [0 to 3] | 0 [0 to 4] | 0 [0 to 4] | 0 [0 to 6]

33. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Titer of 1:40 or Greater
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of subjects with Neut titer >= 1:40 was calculated for each study group from the available results at 7 days post first vaccination (Day 8).
Time Frame: Day 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 103 | 103 | 56
percentage of participants | 0 [0 to 3] | 0 [0 to 4] | 0 [0 to 4] | 0 [0 to 6]

34. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Titer of 1:40 or Greater
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study group from the available results at 21 days post first vaccination (Day 22).
Time Frame: Day 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 104 | 102 | 102 | 56
percentage of participants | 1 [0 to 5] | 0 [0 to 4] | 2 [0 to 7] | 0 [0 to 6]

35. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Titer of 1:40 or Greater
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study group from the available results at 7 days post second vaccination (Day 29).
Time Frame: Day 29
Population: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study group from the available results at 7 days post second vaccination (Day 29).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 96 | 97 | 97 | 54
percentage of participants | 33 [24 to 44] | 29 [20 to 39] | 42 [32 to 53] | 0 [0 to 7]

36. Secondary Outcome: Percentage of Participants Achieving Seroconversion Defined by Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. Day 8 is 7 days after the first dose of H7N9.
Time Frame: Day 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 103 | 103 | 56
percentage of participants | 0 [0 to 3] | 0 [0 to 4] | 2 [0 to 7] | 4 [0 to 12]

37. Secondary Outcome: Percentage of Participants Achieving Seroconversion Defined by Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. Day 22 is 21 days after the first dose of H7N9.
Time Frame: Day 22
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 104 | 102 | 102 | 56
percentage of participants | 4 [1 to 10] | 0 [0 to 4] | 6 [2 to 12] | 4 [0 to 12]

38. Secondary Outcome: Percentage of Participants Achieving Seroconversion Defined by Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and mininmum 4-fold rise in post-vaccination antibody titer. Day 29 is 7 days after the second dose of H7N9.
Time Frame: Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 96 | 97 | 97 | 54
percentage of participants | 34 [25 to 45] | 26 [17 to 36] | 40 [30 to 51] | 2 [0 to 10]

39. Secondary Outcome: Percentage of Participants Achieving Seroconversion Defined by Neutralizing (Neut) Antibodies
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. Day 8 is 7 days after the first dose of H7N9.
Time Frame: Day 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 105 | 103 | 103 | 56
percentage of participants | 0 [0 to 3] | 0 [0 to 4] | 0 [0 to 4] | 0 [0 to 6]

40. Secondary Outcome: Percentage of Participants Achieving Seroconversion Defined by Neutralizing (Neut) Antibodies
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. Day 22 is 21 days after the first dose of H7N9.
Time Frame: Day 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 104 | 102 | 102 | 56
percentage of participants | 1 [0 to 5] | 0 [0 to 4] | 2 [0 to 7] | 0 [0 to 6]

41. Secondary Outcome: Percentage of Participants Achieving Seroconversion Defined by Neutralizing (Neut) Antibodies
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. Day 29 is 7 days after the second dose of H7N9.
Time Frame: Day 29
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
Number analyzed (Participants) | 96 | 97 | 97 | 54
percentage of participants | 33 [24 to 44] | 29 [20 to 39] | 42 [32 to 53] | 0 [0 to 7]

ADVERSE EVENTS:
Time Frame: Solicited events and clinical laboratory evaluations for safety were collected from the time of each study vaccination through 7 days after each study vaccination. Unsolicited non-serious AEs were collected from the time of each study vaccination through approximately 21 days after each study vaccination. SAEs and MAAEs, including NOCMCs and PIMMCs, were collected from the time of the first study vaccination through the final study visit, approximately 12 months after the last study vaccination.
Arm/Group | 3.75 mcg A/H7N9+MF59 | 7.5 mcg A/H7N9+MF59 | 15 mcg A/H7N9+MF59 | 15 mcg A/H7N9
All-Cause Mortality (participants affected / at risk) | 0/105 | 1/105 | 0/104 | 0/57
Serious Adverse Events (participants affected / at risk) | 1/105 | 6/105 | 4/104 | 1/57
Other Adverse Events (participants affected / at risk) | 93/105 | 95/105 | 92/104 | 45/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.75 mcg A/H7N9+MF59 (N=105) | 7.5 mcg A/H7N9+MF59 (N=105) | 15 mcg A/H7N9+MF59 (N=104) | 15 mcg A/H7N9 (N=57)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chlamydial Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anastomotic Ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple Injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.75 mcg A/H7N9+MF59 (N=105) | 7.5 mcg A/H7N9+MF59 (N=105) | 15 mcg A/H7N9+MF59 (N=104) | 15 mcg A/H7N9 (N=57)
Nausea (Gastrointestinal disorders) | 9 (9) | 9 (11) | 13 (13) | 5 (8)
Fatigue (General disorders) | 35 (43) | 33 (41) | 36 (39) | 11 (15)
Feeling Hot (General disorders) | 7 (7) | 6 (6) | 11 (11) | 4 (4)
Malaise (General disorders) | 16 (17) | 21 (24) | 21 (22) | 10 (14)
Upper Respiratory Tract Infection (Infections and infestations) | 11 (12) | 16 (16) | 16 (18) | 5 (6)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Tooth Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Blood Bilirubin Increased (Investigations) | 1 (1) | 2 (3) | 2 (4) | 4 (7)
Hemoglobin Decreased (Investigations) | 6 (11) | 6 (15) | 3 (5) | 9 (12)
Platelet Count Increased (Investigations) | 3 (7) | 4 (9) | 6 (8) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 12 (26) | 9 (11) | 6 (11) | 4 (7)
White Blood Cell Count Increased (Investigations) | 4 (8) | 4 (8) | 6 (8) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6) | 9 (9) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (23) | 23 (28) | 22 (27) | 7 (8)
Headache (Nervous system disorders) | 34 (41) | 31 (39) | 29 (34) | 14 (16)
Injection Site Erythema (General disorders) | 21 (27) | 14 (19) | 13 (17) | 8 (10)
Injection Site Haemorrhage (General disorders) | 4 (4) | 3 (4) | 9 (9) | 4 (4)
Injection Site Induration (General disorders) | 12 (15) | 14 (18) | 14 (16) | 4 (4)
Injection Site Pain (General disorders) | 48 (65) | 43 (60) | 46 (66) | 6 (7)
Injection Site Pain (Tenderness) (General disorders) | 75 (120) | 74 (112) | 71 (108) | 16 (19)
Injection Site Pruritus (General disorders) | 5 (5) | 3 (3) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT03682120/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT03682120/SAP_001.pdf